CLINICAL TRIAL: NCT04335149
Title: 1- Year Follow-up After TAVR Performed Without Systematic Intensive Care Unit Admission
Brief Title: Follow-up After TAVR Without Systematic Intensive Care Unit Admission
Acronym: TAVICU
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0169
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic valve stenosis; TAVI
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COREVALVE: Patients undergoing a TAVI at Montpellier University Hospital since 2017 with implantation of a COREVALVE
- EDWARDS: Patients undergoing a TAVI at Montpellier University Hospital since 2017 with implantation of a EDWARDS

SUMMARY:
Since the first case described in 2002, TAVI (transcatheter Aortic Valve Implantation) revolutionized the management of severe symptomatic aortic stenosis. Initially reserved for patients with prohibitive surgical risk, transfemoral TAVI in now indicated according to European Guidelines for patients at intermediate surgical risk and those > 75 ans. Post-procedure intensive care admission (ICU), initially considered as the rule regarding the risk of complications, (particularly conductive disorders), may be avoided in 1/3 of patients regarding drastic reduction in serious complications and growing experience of operators as the investigator shown in a previous prospective study. Predictive criteria for low-risk of complications were therefore established by our team and may be used in routine to select patients that might avoid ICU. However, long-term impact of this triage strategy remains unknown.

Objective:

The objective of this study is to assess 1-year outcomes according to unit admission selection (ICU or conventional care unit (CCU)) in patients undergoing TAVI.

Since the first case described in 2002, TAVI (transcatheter Aortic Valve Implantation) revolutionized the management of severe symptomatic aortic stenosis. Initially reserved for patients with prohibitive surgical risk, transfemoral TAVI in now indicated according to European Guidelines for patients at intermediate surgical risk and those > 75 ans. Post-procedure intensive care admission (ICU), initially considered as the rule regarding the risk of complications, (particularly conductive disorders), may be avoided in 1/3 of patients regarding drastic reduction in serious complications and growing experience of operators as the investigator shown in a previous prospective study. Predictive criteria for low-risk of complications were therefore established by our team and may be used in routine to select patients that might avoid ICU. However, long-term impact of this triage strategy remains unknown.

Objective:

The objective of this study is to assess 1-year outcomes according to unit admission selection (ICU or conventional care unit (CCU)) in patients undergoing TAVI.

DETAILED DESCRIPTION:
Since the first case described in 2002, indications of TAVI (transcatheter Aortic Valve Implantation) procedures increased in the treatment of symptomatic severe aortic stenosis. Initially reserved for inoperable patients or at high surgical risk, the indication for TAVI was recently extended to patients at intermediate surgical risk. Post-procedure intensive care admission (ICU) was initially considered the rule for all patients regarding the risk of high-grade conductive disorders, vascular or neurological complications. However, given the drastic reduction in serious complications and the increasing number of procedures, systematic ICU admission may be safely avoided. Selection criteria for ICU admission were established by our team in a previous study. The use of these low risk criteria, the growing experience of operators as well as technological improvements allow to safely avoid ICU admission in 1/3 of patients. However, long-term impact of this triage strategy remains unknown.

Objective:

The objective of this study is to assess 1-year outcomes of patients undergoing TAVI according to unit admission (ICU or conventional care unit (CCU)).

Methods This monocentric observational study retrospectively includes all patients undergoing TAVI at the Montpellier University Hospital from 2017. TAVI is indicated in patients with symptomatic severe aortic stenosis with a life expectancy > 1year and contra-indicated for conventional surgery, at high risk or intermediate surgical risk> 75 years after "heart team" decision. Exclusion criteria are patients who died before unit admission or referred a non-cardiological unit after the procedure. Two groups of patients are defined: (1) patients referred to the ICU and (2) patients referred to the CCU after the procedure according to risk-stratification criteria. Low-risk of complications criteria were defined as the absence of major comorbidities, hemodynamic stability, absence of pre-procedure right bundle branch block, LVEF> 40% and absence of procedural complications, particularly the absence of any new conductive disorder after 2 hours monitoring. The primary endpoint is 1-year major events (all-cause mortality, major cardiovascular event and rehospitalization for cardiac causes) according to the VARC-2 criteria. The secondary endpoints include hospitalization duration, 1-month major events and all-cause mortality during follow-up > 1 year depending on the group.

Data assessment Data on patients' baseline characteristics, procedural details and in-hospital outcomes is collected from a prospective TAVI database. No additional testing or biological samples were specifically required for this study

ELIGIBILITY:
Inclusion criteria:

* age > 18 yo
* Patients undergoing a TAVI at Montpellier University Hospital since 2017
* With implantation of a COREVALVE or EDWARDS

Exclusion criteria:

* Minor patient
* Patient unable to give consent for reasons of understanding or language barrier
* Death before unit admission
* Patients referred to a non cardiological unit after the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing TAVI for aortic valve stenosis from January 2017
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Description of causes mortality | 1 year
  All cause mortality
Description of causes heart failure | 1 year
  All cause heart failure
Description of causes rehospitalisation | 1 year
  All cause rehospitalisation

SECONDARY OUTCOMES:
hospitalization duration | 1 month
  hospitalization duration

CONTACTS AND LOCATIONS:
Overall Officials: Florence Leclercq, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC